CLINICAL TRIAL: NCT00130351
Title: A 3-week Multicenter Study Investigating Patient Use and Functionality of Formoterol in a Novel Inhalation Device in Patients With Asthma
Brief Title: A 3-week Study Investigating Patient Use and Functionality of Formoterol in a Novel Inhalation Device in Patients With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CFOR258F2309
Record Dates: First submitted 2005-08-08; First posted 2005-08-15 (Estimated); Last update posted 2023-05-19 (Actual); Status verified 2011-10

CONDITIONS: Asthma
Keywords: asthma, formoterol multi-dose dry powder inhaler (MDDPI)
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Device: formoterol

SUMMARY:
This study is designed to investigate the ability of patients with asthma to properly use a new multi-dose dry powder inhaler (MDDPI) device in a real-life situation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are capable of understanding the directions for device usage, evaluating device function and completing the patient diary
* Patients who have a current diagnosis of asthma
* Patients who have a documented forced expiratory volume at 1 second (FEV1) reversibility of at least 12% over baseline value following administration of a bronchodilator (i.e. "historical" reversibility) or demonstrate a >12% increase in FEV1 over their baseline value within 30 minutes after inhalation of up to 360 µg (4 puffs) of albuterol at Visit 1. The administration of albuterol for the reversibility test must be within 30 minutes after baseline spirometry.

Exclusion Criteria:

* Patients who were enrolled in study CFOR258F2304 or CFOR258F2306, or who have any experience using the Certihaler® device.
* QTc above 450 milliseconds for males and 470 milliseconds for females, or any findings on the screening electrocardiogram (ECG) that in the opinion of the investigator would present a safety hazard for continuation in the study
* Patients who have a known history of untoward reactions to sympathomimetic amines or to inhaled medications or to any of the individual components in those therapies
* Other protocol-defined inclusion and exclusion criteria apply

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2005-07; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Device use: Patients were instructed to record the number appearing in the dose counter window after their dose on the diary card.
Safety: Assessed by adverse events, physical examinations, vital signs abnormalities, forced expiratory volume in 1 second (FEV1) and screening ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (12):
- United States (12):
  - Allergy and Asthma Specialists Medical Group and Research Ct, Huntington Beach, California
  - Allergy and Asthma Medical Group & Research Center, San Diego, California
  - Allergy & Asthma Associates of Santa Clara Res. Center, San Jose, California
  - Colorado Allergy and Asthma Centers, PC, Denver, Colorado
  - Colorado Allergy and Asthma Centers, PC, Englewood, Colorado
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Northeast Medical Research Associates, Inc, North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - The Asthma & Allergy Center, PC, Papillion, Nebraska
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Allergy Associates Research Center, Portland, Oregon